CLINICAL TRIAL: NCT04966689
Title: Comparison of The Effect of Speech Therapy , Music-therapy and Combined Speech and Music Therapy on the Vocal Characteristics of People With PD by Using Telerehabilitation
Brief Title: The Effect of Combined Speech and Music-therapy on the Speech Characteristics of People With Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-06-30; First posted 2021-07-19 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Speech Disorders; Voice Disorders; Parkinson Disease
MeSH Terms: conditions — Speech Disorders; Voice Disorders; Parkinson Disease | interventions — Music Therapy; Speech Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined speech and music therapy (Experimental): the telerehabilitation intervention that include both speech therapy and music therapy at the same time
  Interventions: Behavioral: combined speech and music therapy
- speech therapy (Active Comparator): A behavioural speech therapy program including breathing exercises, loudness, pitch, and intelligibility which are adapted from Lee Silverman Voice Treatment (LSVT) and voice exercises Which is delivered through telerehabilitation
  Interventions: Behavioral: speech therapy
- music therapy (Active Comparator): music exercises Will be designed based on the music therapy protocols of previous studies Which is delivered through telerehabilitation
  Interventions: Behavioral: music therapy

INTERVENTIONS:
Behavioral: combined speech and music therapy — he telerehabilitation intervention that include both speech therapy and music therapy at the same time
  Arms: combined speech and music therapy
Behavioral: speech therapy — A behavioural speech therapy program including breathing exercises, loudness, pitch, and intelligibility which are adapted from Lee Silverman Voice Treatment (LSVT) and voice exercises Which is delivered through telerehabilitation
  Arms: speech therapy
Behavioral: music therapy — music exercises Will be designed based on the music therapy protocols of previous studies Which is delivered through telerehabilitation
  Arms: music therapy

SUMMARY:
Speech and voice disorders are observed in almost 90% of patients with PD during their course of illness. Reduced voice pitch inflections or monotone speech, reduced vocal loudness, prosody disorders, the imprecise articulation of the consonants, hoarseness, and breathy voice is also observed in patients with PD; these symptoms often lead to reduced speech intelligibility. The aim of this study will to investigate the possible changes in the voice and speech features in people with PD after a combined speech and music therapy using Telerehabilitation.

DETAILED DESCRIPTION:
the investigators of this study propose to conduct a pilot randomized, controlled trial in patients with PD to assess the potential effectiveness of a Telerehabilitation intervention that encourage a higher level of speech performance. The investigators hypothesize that patients in the combined treatment group will have more and better improve in the study outcome measures after treatment and 3 month follow up, as compared with patients in speech therapy group and music therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease (IPD)
* Patients who are in stages 1-3 according to Hoehn & Yahr test
* Native language is persian
* The patient or family complains about the person's speech condition
* Adequate vision and hearing
* No history of stroke, head injury, brain surgery, laryngeal diseases such as vocal cord nodules
* No other neurological disorders other than IPD
* Do not use treatment other than medication (such as deep brain stimulation surgery (DBS)
* informed consent

Exclusion Criteria:

* If a patient develops a stroke or other neurological complication during treatment, they are excluded from the treatment
* Lack of cooperation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
loudness | Change from Baseline in loudness at 4 weeks and 3 month follow up
  Change in loudness over the period of the study which will be based on analysis of acoustic recordings. Loudness of voice will be measured in produce the vowel /a /, reading and spontaneous speech. Data will be analyzed using Praat, freeware program for the analysis and reconstruction of acoustic speech signals.

SECONDARY OUTCOMES:
Voice Handicap Index (VHI) | Change from Baseline in VHI at 4 weeks and 3 month follow up
  Change in Persian version of Voice Handicap Index (VHI) over the period of the study. The VHI measures the influence of voice problems on a patient's quality of life. The VHI is a 30 item scale. The total scores range is 0-120. A score 60-120 indicates severe voice problem.
maximum phonation time (MPT) | Change from Baseline in MPT at 4 weeks and 3 month follow up
  Change in maximum phonation time (MPT) over the period of the study. MPT will be measured by asking the subject to produce the long vowel /a/. This vocalization is measured three times, and the longest MPT is recorded.
Speech Intelligibility | Change from Baseline in Speech Intelligibility at 4 weeks and 3 month follow up
  Change in fudalla speech intelligibility rating scale over the period of the study. This scale consists of 7 rates in which the number 1 indicates Speech is not intelligible and number 7 indicates Speech is totally intelligible.
Swallowing Disturbance Questionnaire (SDQ) | Change from Baseline in SDQ at 4 weeks and 3 month follow up
  Change in Persian version of Swallowing Disturbance Questionnaire (SDQ) over the period of the study. The SDQ is a 15 item scale. The total scores range is 0-45. A score higher 11 indicates swallowing difficulty.
Dysphagia handicap index (DHI) | Change from Baseline in DHI at 4 weeks and 3 month follow up
  Change in Persian version of Dysphagia handicap index (DHI) over the period of the study. The DHI is one of the instruments used for measuring a dysphagic patient's self-assessment. it reflects the patient's quality of life. DHI is a 25 item scale. The total scores range is 0-100. A higher score indicates a greater impact of swallowing disorders on quality of life
northwest dysphagia patient check sheet (NDPCS) | Change from Baseline in NDPCS at 4 weeks and 3 month follow up
  Change in Persian version of northwest dysphagia patient check sheet (NPCS) scores over the period of the study. The NDPCS has five and 28 items. Each item is scored as safe or unsafe. The total score is calculated from the total number of unsafe items. The more unsafe observations indicates swallowing difficulty.
Geriatric Depressive Scale (GDS) | Change from Baseline in GDS at 4 weeks and 3 month follow up
  Change in Persian version of Geriatric Depressive Scale (GDS) scores over the period of the study. GDS is a 15 item scale. Each item is scored as yes or no. More than 5 signs indicate the possibility of depression and more than 10 signs of depression indicate definite depression.
quality of life (QoL) | Change from Baseline in QOL at 4 weeks and 3 month follow up
  Change in SF-36 questionnaire over the period of the study. Quality of life will be measured using SF-36 questionnaire. SF-36 is a 36 item scale. The total scores range is 0-100. A higher score indicates a better quality of life.
jitter | Change from Baseline in jitter at 4 weeks and 3 month follow up
  Change in jitter over the period of the study, which will be based on analysis of acoustic recordings. jitter will be measured in produce the vowel /a/. Data will be analyzed using Praat, freeware program for the analysis and reconstruction of acoustic speech signals.
shimmer | Change from Baseline in shimmer at 4 weeks and 3 month follow up
  Change in shimmer over the period of the study, which will be based on analysis of acoustic recordings. shimmer will be measured in produce the vowel /a/. Data will be analyzed using Praat, freeware program for the analysis and reconstruction of acoustic speech signals.
highest and lowest frequency | Change from highest and lowest frequency at 4 weeks and 3 month follow up
  Change in highest and lowest frequency over the period of the study, which will be based on analysis of acoustic recordings. highest and lowest frequency will be measured by asking the subject to produce the vowel /a/ as high and low frequency as they can produces. Data will be analyzed using Praat, freeware program for the analysis and reconstruction of acoustic speech signals.

CONTACTS AND LOCATIONS:
Overall Officials: Reyhaneh Mohammadi, Study Director — Iran university of medical science
Locations (1):
- Iran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohseni Z, Mohamadi R, Habibi SAH, Saffarian A, Abolghasemi J. Voice improvement following conventional speech therapy combined with singing intervention in people with Parkinson's disease: A three-arm randomised controlled trial. Int J Lang Commun Disord. 2023 Sep-Oct;58(5):1752-1767. doi: 10.1111/1460-6984.12900. Epub 2023 Jun 7. PMID 37282797